CLINICAL TRIAL: NCT00740467
Title: Allograft of Hematopoietic Stem Cells With Reduced-intensity Conditioning From a HLA-haploidentical Family Donor: Phase II Study of Combined Immunosuppression Before and After Transplantation
Brief Title: Stem Cell Transplant in Treating Patients With Hematological Cancer or Other Disorders
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Paoli-Calmettes (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000592923; IPC-ITT-06-01; INCA-RECF0627; EUDRACT-2006-001369-14
Record Dates: First submitted 2008-08-22; First posted 2008-08-25 (Estimated); Last update posted 2010-01-28 (Estimated); Status verified 2009-07

CONDITIONS: Graft Versus Host Disease; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Precancerous Condition
Keywords: graft versus host disease; adult acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); recurrent adult acute myeloid leukemia; adult acute lymphoblastic leukemia in remission; recurrent adult acute lymphoblastic leukemia; accelerated phase chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; refractory multiple myeloma; relapsing chronic myelogenous leukemia; recurrent adult Hodgkin lymphoma; adult nasal type extranodal NK/T-cell lymphoma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult grade III lymphomatoid granulomatosis; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult T-cell leukemia/lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent grade I lymphomatoid granulomatosis; recurrent grade II lymphomatoid granulomatosis; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; splenic marginal zone lymphoma; refractory chronic lymphocytic leukemia
MeSH Terms: conditions — Graft vs Host Disease; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Precancerous Conditions; Congenital Abnormalities; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myeloid, Chronic-Phase; Hodgkin Disease; Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Antilymphocyte Serum; Busulfan; Cyclophosphamide; Cyclosporine; fludarabine phosphate; Mycophenolic Acid

INTERVENTIONS:
Biological: anti-thymocyte globulin
Drug: busulfan
Drug: cyclophosphamide
Drug: cyclosporine
Drug: fludarabine phosphate
Drug: mycophenolate mofetil
Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation

SUMMARY:
RATIONALE: Giving chemotherapy, such as fludarabine, busulfan, and cyclophosphamide, together with antithymocyte globulin before a donor stem cell transplant helps stop the growth of cancer and abnormal cells. Giving chemotherapy before or after transplant also stops the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer and abnormal cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving cyclosporine and mycophenolate mofetil after the transplant may stop this from happening.

PURPOSE: This phase II trial is studying how well stem cell transplant works in treating patients with hematological cancer or other disorders.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the incidence of graft acceptance in patients with hematological disorders treated with combined immunosuppression before and after HLA-haploidentical hematopoietic stem cell transplantation.

Secondary

* Evaluate efficacy of this regimen in these patients.
* Evaluate toxicity of this regimen in these patients.
* Assess survival of patients treated with this regimen.

OUTLINE: This is a multicenter study.

* Reduced-intensity conditioning: Patients receive fludarabine phosphate IV on days -6 to -1, busulfan IV on days -6 to -5, and anti-thymocyte globulin IV on days -4 to -1.
* Transplantation: Patients undergo transplantation of donor hematopoietic stem cells on day 0. Patients also receive cyclophosphamide IV on day 3 and filgrastim (G-CSF) beginning on day 4 and continuing until blood counts recover.
* Immunosuppression: Patients receive cyclosporine IV beginning on day -2 and continuing for 6 months and mycophenolate mofetil 4 times a day on days 4-84.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of any of the following hematological cancers with a poor prognosis:

  * Acute myeloid leukemia meeting 1 of the following criteria:

    * Third complete remission (CR3) or beyond
    * CR2 after an early bone marrow relapse (< 24 months)
    * Refractory disease after ≥ 2 chemotherapy courses of induction therapy
  * Acute lymphoblastic leukemia meeting 1 of the following criteria:

    * CR3 after ≥ 1 bone marrow relapse
    * CR2 after early bone marrow relapse (currently or within 6 months after stopping maintenance therapy)
  * Chronic myelogenous leukemia meeting the following criteria:

    * Accelerated phase
    * Second chronic phase
    * No other treatment options
  * Multiple myeloma meeting the following criteria:

    * Failed conventional therapy (including autologous hematopoietic stem cell transplantation)
    * No other treatment alternatives
  * Chronic lymphocytic leukemia meeting the following criteria:

    * Failed conventional therapy
    * No other treatment alternatives
  * Hodgkin lymphoma meeting the following criteria:

    * Failed conventional therapy
    * No other treatment alternatives
  * Non-Hodgkin lymphoma meeting the following criteria:

    * Failed conventional therapy
    * No other treatment alternatives
* Not eligible for standard myeloablative allograft due to increased toxicity
* Healthy related donor available and meeting the following criteria:

  * Brother, sister, father, mother, cousin, uncle, or aunt
  * At least an identical HLA haplotype

    * Identical genotype on 1 haplotype (in terms of HLA-A, B, C, and DR)
    * Different on ≤ 4 alleles on the other haplotype
* No HLA-identical intra- or extra-familial donor cord blood available within the next 3 months

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No contraindication to allogeneic transplantation, including any of the following:

  * Cardiac systolic ejection fraction < 40%
  * DLCO level limiting use of fludarabine
  * Creatinine clearance < 30 mL/min
  * Transaminases and/or bilirubin > 3 times upper limit of normal (unless due to Gilbert disease or cancer)
  * HIV seropositivity
  * Human T-cell lymphotrophic virus type 1 seropositivity
  * Uncontrolled bacterial, viral, or fungal infection
* No contraindication to any of the study drugs
* No prior or concurrent psychiatric illness
* No other cancer in the past 5 years except for basal cell skin cancer or carcinoma in situ of the cervix
* No concurrent serious, uncontrolled condition
* No patients deprived of liberty or subject to legal protection

PRIOR CONCURRENT THERAPY:

* No participation in a study of allografts in the past month

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-01; Primary Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of graft acceptance

CONTACTS AND LOCATIONS:
Overall Officials: Didier Blaise, MD, Study Chair — Institut Paoli-Calmettes
Locations (1):
- Marseille Institute of Cancer - Institut J. Paoli and I. Calmettes, Marseille, France